CLINICAL TRIAL: NCT00375882
Title: Mild Hypothermia During Cochlear Implantation
Brief Title: Safety Study to Evaluate the Effect of Lowering Body Temperature During Cochlear Implantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: as specified in the protocol
Sponsor: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20060088
Record Dates: First submitted 2006-09-11; First posted 2006-09-13 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Hypothermia
MeSH Terms: conditions — Hypothermia | interventions — Cochlear Implantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cochlear implantation with mild hypothermia (Other)
  Interventions: Procedure: hypothermia; Procedure: cochlear implantation with mild hypothermia

INTERVENTIONS:
Procedure: hypothermia
Procedure: cochlear implantation with mild hypothermia

SUMMARY:
Hypothesis: Mild Hypothermia has a protective effect on residual hearing of patients undergoing cochlear implantation

DETAILED DESCRIPTION:
Hypothermia has been shown to have a protective effect following trauma to the central nervous system and the peripheral auditory system. We have previously demonstrated a protective effect of mild hypothermia on auditory function caused by cochlear implant electrodes in animal models. Preservation of residual hearing of patients undergoing cochlear implantation is highly desirable and based on these animal studies, it may be possible to achieve in human subjects using mild degrees of hypothermia. We propose to investigate the hypothesized protective effect of intra-operative hypothermia on adult subjects undergoing cochlear implantation.

Inclusion Criteria: Adults greater than or equal to 18 years of age with some measurable auditory function who are undergoing cochlear implantation as routine management of severe to profound hearing loss.

Exclusion Criteria: Pure tone average hearing (mean of .5, 1 and 2 KHz) worse than 100dB; Age > 70 years; History of arrhythmia or ischemic heart disease; sickle cell trait or disease; immune incompetence; coagulation disorders; revision cochlear implant; body-mass index > 35; cold related disorders.

Phase I: Up to 40 healthy adult subjects who have qualified for CI will undergo implantation with core body temperature lowered to 34 degree Centigrade for approximately one hour before electrode insertion and 30 minutes after insertion. Otherwise, the surgical technique will be unchanged from our standard procedure.

The heating/cooling blanket is an FDA approved device. similar temperature controlling blankets are used in virtually all operations done under general anesthesia. Each subject's temperature will be gradually lowered only after they are put to sleep. Warming will being at least 30 minutes before the subject is awakened. We will measure and record the subject's temperature every 5 to 15 minutes while they are in the operating room and also while they are in the recovery room.

Each subject will undergo a battery of audiometric tests (CNC words, HINT sentences, pure tone thresholds, and immittance) within one month prior to implantation, at one month post operatively, at 6 months post operatively and 1 year postoperatively. Outcomes will be analyzed by PI after 10 subjects have completed the 1 month test interval. If outcomes indicate proof of principle (measurable pure tone responses in greater than or equal to 60% of subjects), phase two of the study will be initiated. If not, outcomes will be analyzed after 20, 30, and 40 subjects until evidence of hearing conservation or lack of it is established, leading to the following study or precluding it.

Phase II: Up to 80 healthy adults who have qualified for CI will be randomized into control group (CI surgery using standard procedure at core body temperature of 37 degree C) or active group (identical core body temperature of 34 degrees C). Subjects will be randomized using a random table of numbers. The patient, surgeon and audiologist will be blinded to the group assignment. Only the study coordinator will have the sequestered and locked list of randomization and blinding. Only the anesthesiologist will know the patients' assignment at the time of surgery. The audiologist will not be present in the O.R. or in the outpatient clinic, but will only test the patient post surgery. Each subject will undergo a battery of audiometric tests (CNC words, HINT sentences, pure tone thresholds, and immittance) just prior to implantation, at 1 month post operatively, at 6 months post operatively and at 1 year postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Adults undergoing measurable auditory function who are undergoing cochlear implantation as routine management of severe to profound hearing loss.

Exclusion Criteria:

* Pure tone average hearing ( mean of .5, 1 adn 2 KHz) worse than 100dB
* Age> 70 years
* History of arrhythmia or ischemic heart disease
* Sickle cell trait or disease
* Immune incompetence; coagulation disorders
* Revision cochlear implant; body-mass index >35
* Cold related disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-03; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
To determine if mild hypothermia has a protective effect on residual hearing of patients undergoing cochlear implantation. | one month post cochlear implantation

SECONDARY OUTCOMES:
To determine if mild hypothermia has a protective effect on residual hearing of patients undergoing cochlear implantation | one year post cochlear implantation

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Balkany, M.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miller School of Medicine, Ear Institute, Miami, Florida, United States